CLINICAL TRIAL: NCT03295643
Title: Outcomes From a Mobile Smoking Cessation Program During a Monitoring Period of 6 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Marler, MD (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Marler, MD, Senior Director, Clinical and Medical Affairs, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-601
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: All subjects experience same program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mobile smoking cessation program (Other): Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
  Interventions: Device: Mobile smoking cessation program and CO breath sensor device

INTERVENTIONS:
Device: Mobile smoking cessation program and CO breath sensor device — Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.

SUMMARY:
Prospective, open label, single center clinical study enrolling 260 subjects in a mobile smoking cessation program using a smartphone app and a handheld breath sensor with coaching support over a six month period.

DETAILED DESCRIPTION:
This is a prospective, open label, single center clinical study enrolling 260 subjects in a mobile smoking cessation program using a smartphone app and handheld breath sensor with coaching support over a six month period. Measurements include user engagement and retention in the program, attitude towards smoking and smoking behavior, quit rates, relapse rates, and quality of life over the study period, as well as user feedback on the program.

Potential participants will complete an online screening form. Eligible participants will be called to confirm eligibility, discuss the study, and have their questions about the study answered. Interested eligible participants will then be emailed the registration link, which includes the electronic informed consent. After providing electronic informed consent, subjects register online and receive the hand held device which measures carbon monoxide (CO) which correlates to smoking behavior.

Baseline questionnaires (demographics, smoking history, and attitude towards smoking) are completed, and subjects then self-train to use the breath sensor and smartphone app and allows viewing of CO sample values. The app also provides the user with ability to log cigarettes, view cigarette consumption trends, view instructional videos, complete educational activities and challenges, and engage with a coach.

Participants will experience the program in 5 phases and then complete the study at approximately six months after enrolling,activating device and app.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* English speaking
* Smokes daily
* Smokes 5 or more cigarettes per day
* Owns and uses a smartphone (iPhone 5 and above, operating system iOS 9.0 and above, or, Android 4.4 and above, operating system Android 4.4 and above)
* Employed at least 20 hours per week
* Lives in the USA
* Understands and willing to sign the Informed Consent Form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Utley, MD, Principal Investigator — Pivot Health Technologies, Inc (formerly Carrot Sense)
Locations (1):
- Carrot Inc., Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marler JD, Fujii CA, Galanko JA, Balbierz DJ, Utley DS. Durability of Abstinence After Completing a Comprehensive Digital Smoking Cessation Program Incorporating a Mobile App, Breath Sensor, and Coaching: Cohort Study. J Med Internet Res. 2021 Feb 15;23(2):e25578. doi: 10.2196/25578. PMID 33482628
- [Derived] Marler JD, Fujii CA, Utley DS, Tesfamariam LJ, Galanko JA, Patrick H. Initial Assessment of a Comprehensive Digital Smoking Cessation Program That Incorporates a Mobile App, Breath Sensor, and Coaching: Cohort Study. JMIR Mhealth Uhealth. 2019 Feb 4;7(2):e12609. doi: 10.2196/12609. PMID 30670372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Online recruitment
Pre-assignment Details: Phone call to confirm eligibility.
Groups:
- Mobile Smoking Cessation Program: Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
  Mobile smoking cessation program and CO breath sensor device: Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
  The mobile smoking cessation program includes 5 phases with the following names and timelines:
  Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days. Quit = 7 days. Secure = 11 weeks.
Period: Overall Study
Arm/Group | Mobile Smoking Cessation Program
Started | 319
Completed Explore Stage | 283
Completed Build Stage | 183
Completed Mobilize Stage | 139
Completed Quit Stage | 131
Completed Secure Stage | 126
Completed (Completed the end-of-Pivot questionnaire and thus completed the study) | 272
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184
  Male | 135
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 264
  Ethnicity: African American | 22
  Ethnicity: Hispanic | 15
  Ethnicity: Asian | 5
  Ethnicity: American Indian or Alaska Native | 4
  Ethnicity: Native Hawaiian or other Pacific Islander | 2
  Ethnicity: Other | 7
Region of Enrollment [Number; unit: participants]
  United States | 319
Cigarettes smoked per day [Mean (Standard Deviation); unit: Cigarettes per day] | 17.7 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Explore Stage
Description: For the number of participants who started the Explore Stage, the proportion who completed the Explore Stage.
Time Frame: Assessment at the end of the Explore stage; 9 days after activating the app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 283

2. Primary Outcome: Number of Participants Who Completed the Build Stage
Description: For the number of participants who started the Build Stage, the proportion who completed the Build Stage.
Time Frame: Assessment at the end of the Build stage; between 10 and 37 days after activating the app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 183

3. Primary Outcome: Number of Participants Who Completed the Mobilize Stage
Description: For the number of participants who started the Mobilize Stage, the proportion who completed the Mobilize Stage.
Time Frame: Assessment at the end of the Mobilize stage; between 17 and 44 days after activating the app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 139

4. Primary Outcome: Number of Participants Who Completed the Quit Stage
Description: For the number of participants who started the Quit Stage, the proportion who completed the Quit Stage.
Time Frame: Assessment at the end of the Quit Stage; between 24 and 51 days after activating the app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days. Quit = 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 131

5. Primary Outcome: Number of Participants Who Completed the Secure Stage
Description: For the number of participants who started the Secure Stage, the proportion who completed the Secure Stage.
Time Frame: Assessment at the end of the Secure Stage; between 101 and 128 days after activating the app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days. Quit = 7 days. Secure = 11 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 126

6. Secondary Outcome: Readiness to Quit and Goals Related to Smoking Behavior
Description: Are you seriously thinking of quitting smoking? (stage of change) "Yes, within the next 30 days". "Yes, within the next 6 months". "No, not thinking of quitting".
Time Frame: Assessment at the end of the Explore stage; 9 days after activating app and device. Explore = 9 days. Build = 1 day to 4 weeks. Mobilize = 7 days.
Population: Participants who provided baseline and explore stage results
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 281
Participants
  Baseline - Stage of Change: Yes, within the next 30 days | 94
  Baseline - Stage of Change: Yes, within the next 6 months | 176
  Baseline - Stage of Change: No, not thinking of quitting | 11
  End of Explore Stage - Stage of Change: Yes, within the next 30 days | 157
  End of Explore Stage - Stage of Change: Yes, within the next 6 months | 114
  End of Explore Stage - Stage of Change: No, not thinking of quitting | 10

7. Secondary Outcome: Average Percentage Change in Cigarettes Per Day (CPD) by the Pre-Quit Stage
Description: Average percentage change in cigarettes per day (CPD) by the Pre-Quit Stage using repeated measures linear mixed model analysis.
  Model uses all available data on CPD to estimate an average. The Pre-Quit Stage is defined as from the start of the study (activation of the app and device/ Baseline) to the end of the Mobilize Stage.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in cpd
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
percentage change in cpd | -44.5 (3)

8. Secondary Outcome: Weeks of Active Engagement
Description: Engagement defined as interaction with the program at least once within app (app open, daily check-in, responds to coach, logs cigarettes, etc)
  Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
  Mobile smoking cessation program and CO breath sensor device: Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- All Participants: Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
  Mobile smoking cessation program and CO breath sensor device: Mobile smoking cessation program delivered through an app with access to a breath sensor device and coaching support.
Arm/Group | All Participants
Number analyzed (Participants) | 319
weeks | 12.4 (7.1)

9. Secondary Outcome: Number of Participants Who Completed the Program
Description: The number of participants who completed the quit-smoking program.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
Participants | 272

10. Secondary Outcome: Quit Attempts
Description: Number attempt to quit by participant
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 272
quit attempts | 2.4 (3.1)

11. Secondary Outcome: Quit Rate 7-day Point Prevalence
Description: Number of participant who have not smoked in last 7 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 272
Participants | 102

12. Secondary Outcome: Quit Rate 30-day Point Prevalence
Description: Number of participant who have not smoked in last 30 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 272
Participants | 88

13. Secondary Outcome: Number of Participants Who Reported Pivot Increased Their Motivation to Stop Smoking
Description: the number of participants who reported Pivot program (app, breath sensor, and coaching) increased their motivation to stop smoking
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 272
Participants | 233

14. Secondary Outcome: Confidence to Quit
Description: Confidence to quit. Estimate of means and standard errors based on linear mixed model.
  Participants were asked: "If you were to quit smoking right now, how successful would you be?" Answered on a scale from 1 to 10 (1=not at all successful, 10=completely successful).
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
score on a scale
  Baseline Confidence to Quit | 4.2 (0.1443)
  End of Explore Confidence to Quit | 5.9 (0.1508)
  End of Build Confidence to Quit | 6.4 (0.1782)
  End of Mobilize Confidence to Quit | 7.4 (0.1916)

15. Secondary Outcome: Difficulty Maintaining Quit
Description: Difficulty maintaining quit. Estimate of means and standard errors based on linear mixed model.
  Participants were asked: "If you were to quit smoking right now, how difficult do you think it would be to stay smoke-free?" Answered on a scale from 1 to 10 (1=really hard to stay quit, 10=really easy to stay quit).
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile Smoking Cessation Program
Number analyzed (Participants) | 319
score on a scale
  Baseline difficulty maintaining quit | 3.1 (0.1449)
  End of Explore difficulty maintaining quit | 4.9 (0.1531)
  End of Build difficulty maintaining quit | 5.7 (0.1891)
  End of Mobilize difficulty maintaining quit | 6.8 (0.2055)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mobile Smoking Cessation Program
All-Cause Mortality (participants affected / at risk) | 0/319
Serious Adverse Events (participants affected / at risk) | 0/319
Other Adverse Events (participants affected / at risk) | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03295643/Prot_SAP_001.pdf